CLINICAL TRIAL: NCT05308940
Title: A Phase 1, Single and Multiple Subcutaneous Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics of TB001 Injection in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics of TB001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Turier Biotech Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TB001CT0001
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single-dose of TB001 (Experimental): In the SAD stage, participants will receive subcutaneous injection of TB001 once on Day 1, planning to ascend from 20 μg, 60 μg，150 μg，300 μg，600μg to 900 μg or higher dose (whether to proceed to the next higher cohort based on dose escalation criteria). Actual dose of TB001 may vary based on safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TB001
- Multiple-dose of TB001 (Experimental): In the MAD stage, participants will receive subcutaneous injection of TB001 once daily for 7 days, planning to ascend from 60 μg，150ug to 300 μg or higher dose (whether to proceed to the next higher cohort based on dose escalation criteria). Actual dose of TB001 may vary based on safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TB001
- Single-dose of placebo (Placebo Comparator): In the SAD stage, participants will receive subcutaneous injection of placebo once on Day 1.
  Interventions: Drug: Placebo
- Multiple-dose of placebo (Placebo Comparator): In the MAD stage, participants will receive subcutaneous injection of placebo once daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TB001 — once-daily subcutaneous injection, on Day 1 in SAD stage
  Arms: Single-dose of TB001
Drug: TB001 — once-daily subcutaneous injection, on Days 1-7 in MAD stage
  Arms: Multiple-dose of TB001
Drug: Placebo — once-daily subcutaneous injection, on Day 1 in SAD stage
  Arms: Single-dose of placebo
Drug: Placebo — once-daily subcutaneous injection, on Days 1-7 in MAD stage
  Arms: Multiple-dose of placebo

SUMMARY:
It was a randomized, double-blind, placebo-controlled combined single ascending dose (SAD) and multiple ascending dose (MAD) study, evaluating the safety, tolerability and pharmacokinetics of TB001 after single and multiple subcutaneous injections in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Aged 18-55 years (inclusive), male or female.
3. BMI within 18.0-28.0 kg/m2 (inclusive).
4. Have physically and psychologically health judged by the investigator based on the medical history, physical examination, laboratory evaluation, electrocardiogram, etc.
5. Have agreed to take effective contraception measures.

Exclusion Criteria:

1. Have any prior clinically serious disease of any system.
2. Known or suspected allergy to the study drug or any of its ingredients.
3. Severe infection, severe trauma or major surgical operation within 3 months prior to the first administration.
4. History of recurrent or chronic infection within 6 months prior to the first administration.
5. Unable to comply with dietary management during the study period.
6. Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Day 1 and up to Day 28
  An AE is any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship.

SECONDARY OUTCOMES:
Pharmacokinetics exposure of TB001 in SAD and MAD stage | Day 1 , Day 7
  Serum concentrations of TB001 at different timepoints before and after TB001 administration.
Observed immunogenicity of TB001 in MAD stage | Day 1, Day 7, Day 14, Day 28
  Number of subjects who develop detectable ADAs and NAb after TB001 administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Turier Biotech Co., Ltd., Shenzhen, Guangdong, China